CLINICAL TRIAL: NCT03721419
Title: Low-Flow (LF) Oxygen Versus Heated Humidified High-Flow (HF) Therapy Following Tracheostomy
Brief Title: High-Flow Oxygen Therapy Following Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Peggy Watts, Manager, Respiratory Therapy, Barnes-Jewish Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201707165
Record Dates: First submitted 2018-03-29; First posted 2018-10-26 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2019-07

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Intervention Model Description: Crossover study between 2 medical ICUs and 1 Surgical ICU. Patients in one unit will start off with Low Flow (LF) while the other unit will start off with High Flow (HF). After one half of the required sample size is accrued we will crossover the Medicine ICUs with the Surgical ICU.
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- High Flow High Humidity device (Experimental): High Flow High Humidity device arm subjects will be placed on a High Flow Airvo device post tracheostomy with oxygen bled into system which maintains a safe level of patient blood oxygen. This device has its own flow generator built in.
  Interventions: Device: High Flow High Humidity device
- Low Flow High Humidity Device (Active Comparator): Low Flow High Humidity device arm patients will be placed on a Low Flow device post tracheostomy with oxygen bled into system which maintains a safe level of patient blood oxygen.
  Interventions: Device: Low Flow High Humidity device

INTERVENTIONS:
Device: High Flow High Humidity device — High Flow High Humidity device has a flow generator built into the body of unit and can deliver flows between 10 to 60 Liters per minute (LPM) with oxygen bled in as needed in order to deliver specified Fraction of inspired Oxygen (FiO2)
  Other Names: Airvo high flow device
  Arms: High Flow High Humidity device
Device: Low Flow High Humidity device — Standard high humidity trach collar utilizing venturi device bleed in
  Other Names: High Humidity Trach Collar
  Arms: Low Flow High Humidity Device

SUMMARY:
Respiratory failure patients sometimes receive tracheostomy due to difficulty weaning from mechanical ventilation. Efforts to wean patients with a tracheostomy usually involve the administration of oxygen via High Humidity device. There are two major ways of administering oxygen to patients which include low flow delivered at less than 10Liters per minute (LPM) and high-flow delivered at greater than 10LPM. There is not a currently accepted standard of care practice for how to administer oxygen therapy to these patients. Both Low and High Flow are accepted practices in the US.

DETAILED DESCRIPTION:
Many patients with Respiratory Failure undergo tracheostomy due to difficulty weaning from mechanical ventilation. A component of weaning a patient with tracheostomy usually involves the administration of oxygen via High Humidity device. There are two major ways of administering oxygen via High Humidity to patients. They include low flow high humidity; delivered at less than or equal to 10LPM or high-flow humidity, delivered at greater than 10LPM. There is not a currently accepted standard of practice for how to administer oxygen high humidity to patients who receive a tracheostomy due to respiratory failure. Both Low and High Flow high humidity devices are used routinely by health care facilities nationwide. Therefore, the investigators plan to perform a crossover study in both a medicine and surgical Intensive Care Unit to determine which type of oxygen High Humidity therapy should be preferentially utilized. Patients in one Intensive Care Unit will start off with Low Flow high humidity while the alternate unit will start with Hi Flow high humidity. After one half of the required sample size is accrued the investigators will cross over the two ICUs to the alternate type of oxygen High Humidity device. No other respiratory practices will change during the conduct of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients who receive tracheostomy

Exclusion Criteria:

* Non-English speaking and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Days of Mechanical Ventilation (MV) | an average of 1 year
  Time in days from initiation of MV until discontinuance of MV

SECONDARY OUTCOMES:
Days of ICU Stay | an average of 1 year
  The number of days the subject is in the ICU
Days of hospital stay | an average of 1 year
  Time in days from admission to hospital until discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrer M, Sellares J, Valencia M, Carrillo A, Gonzalez G, Badia JR, Nicolas JM, Torres A. Non-invasive ventilation after extubation in hypercapnic patients with chronic respiratory disorders: randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1082-8. doi: 10.1016/S0140-6736(09)61038-2. Epub 2009 Aug 12. PMID 19682735
- [Background] Jaber S, Jung B, Chanques G, Bonnet F, Marret E. Effects of steroids on reintubation and post-extubation stridor in adults: meta-analysis of randomised controlled trials. Crit Care. 2009;13(2):R49. doi: 10.1186/cc7772. Epub 2009 Apr 3. PMID 19344515
- [Background] Glossop AJ, Shephard N, Bryden DC, Mills GH. Non-invasive ventilation for weaning, avoiding reintubation after extubation and in the postoperative period: a meta-analysis. Br J Anaesth. 2012 Sep;109(3):305-14. doi: 10.1093/bja/aes270. PMID 22879654
- [Background] Ferrer M, Valencia M, Nicolas JM, Bernadich O, Badia JR, Torres A. Early noninvasive ventilation averts extubation failure in patients at risk: a randomized trial. Am J Respir Crit Care Med. 2006 Jan 15;173(2):164-70. doi: 10.1164/rccm.200505-718OC. Epub 2005 Oct 13. PMID 16224108
- [Background] Nava S, Gregoretti C, Fanfulla F, Squadrone E, Grassi M, Carlucci A, Beltrame F, Navalesi P. Noninvasive ventilation to prevent respiratory failure after extubation in high-risk patients. Crit Care Med. 2005 Nov;33(11):2465-70. doi: 10.1097/01.ccm.0000186416.44752.72. PMID 16276167